CLINICAL TRIAL: NCT00111852
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Single Bolus, Multinational, Multi-center, Parallel Group, Dose-ranging Study of Desmoteplase (INN) in the Indication of Acute Stroke
Brief Title: Study of Desmoteplase (International Nonproprietary Name [INN]) in Acute Ischemic Stroke (DIAS-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSP-MD-01
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Stroke, Acute
Keywords: Desmoteplase; Acute Ischemic Stroke; Stroke, Acute
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — salivary plasminogen activator alpha 1, Desmodus rotundus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desmoteplase, low dose (Experimental): Desmoteplase 90 mcg/kg, intravenous administration.
  Interventions: Drug: Desmoteplase
- Desmoteplase, high dose (Experimental): Desmoteplase 125 mcg/kg, intravenous administration.
  Interventions: Drug: Desmoteplase
- Placebo (Placebo Comparator): Dose-Match Placebo, intravenous administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmoteplase — Desmoteplase 90 mcg/kg, intravenous administration.
  Arms: Desmoteplase, low dose
Drug: Desmoteplase — Desmoteplase 125 mcg/kg, intravenous administration.
  Arms: Desmoteplase, high dose
Drug: Placebo — Dose-Match Placebo, intravenous administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate desmoteplase (which is a manufactured protein derived from the saliva of the vampire bat) in dissolving clots that are blocking the flow of blood through one (or more) of the blood vessels supplying the brain, thereby reopening the blocked blood vessel and allowing blood to flow again in individuals suffering from ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for study treatment within 3-9 hours after onset of stroke symptoms.
* Score of 4-24 on the NIHSS with clinical signs of hemispheric infarction (i.e. hemiparesis) suggestive of ischemic stroke.

Inclusion Criteria from diagnostic imaging screening:

* Distinct penumbra (at least 20%), measured by MRI (PWI/DWI) or perfusion CT, related to middle cerebral artery (MCA), anterior cerebral artery (ACA), or posterior cerebral artery (PCA) territory in a hemispheric distribution.

Exclusion Criteria:

* History or clinical presentation of intracranial hemorrhage (ICH), subarachnoid hemorrhage, arteriovenous malformation, aneurysm, or cerebral neoplasm.
* Rapidly improving neurological symptoms.
* Pre-stroke MRS score of > 1 (including previous disability).
* Suspected acute vertebral or basilar artery occlusion.
* Current use of anticoagulants and a prolonged prothrombin time.
* Uncontrolled hypertension.
* Baseline hematocrit of < 0.25.
* Baseline platelet count < 100,000/mm3.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | Change from Baseline to day 90
  Improvement of greater than or equal to 8 points from baseline, or NIHSS score less than or equal to 1. The NIHSS score ranges from 0 (least severe) to 42 (more severe).
Modified Rankin Scale (MRS) | Day 90
  Improvement on the Modified Rankin Scale, defined as a score of 0-2. The MRS ranges in severity from 0 (no symptoms) to 6 (Dead).
Barthel Index (BI) score of 75-100. | Day 90
  The Barthel Index (BI) is a scale used to measure performance in basic Activities of Daily Livingranges from 0 (most disablility) to 100 (no disability)

SECONDARY OUTCOMES:
Percentage of patients with improvement in NIHSS score | From Baseline to Day 90
  Improvement of greater than or equal to 8 points from baseline on the NIHSS score, or NIHSS score less than or equal to 1.
Percentage of patients with MRS score of 0-2 | Day 90
Percentage of patients with BI score of 75-100 | Day 90
Infarct Volume | Change from baseline to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lipka, MD, Study Director — Forest Laboratories
Locations (44):
- United States (28):
  - Alabama Neurological Institute, Dept. of Neurology, Birmingham, Alabama
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Brain Matters, Inc., Delray Beach, Florida
  - Melbourne Internal Medicine Associates (MIMA), Melbourne, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Tampa General Hospital, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Indiana Neuroscience Institute, Indianapolis, Indiana
  - Jewish Hospital Healthcare Services, Inc., Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Nevada Neurosciences Institute at Sunrise, Las Vegas, Nevada
  - JFK Medical Center, Edison, New Jersey
  - Presbyterian Hospital, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Erlanger Health System, Chattanooga, Tennessee
  - University of Tennessee, College of Medicine, Chattanooga, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center at Dallas, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Winchester Medical Center, Winchester, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (3):
  - John Hunter Hospital, New Lambton Heights
  - Box Hill Hospital, Victoria
  - Queen Elizabeth Hospital, Woodville
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Leopold-Franzens-Universitat Innsbruck, Innsbruck
  - O O Landesnervenklinik Wagner-Jauregg, Linz
- Canada (2):
  - Walter Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
- Germany (3):
  - Neurologische Universitatsklinik, Bonn
  - Klinik und Poliklinik der Universitat Leipzig, Leipzig
  - Neurologische Klinik Universitat Ulm, Ulm
- University Hospital Amsterdam Department Neurology, Amsterdam, Netherlands
- Spain (2):
  - University Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Doctor Josep Trueta, Girona

REFERENCES:
- [Derived] Warach S, Al-Rawi Y, Furlan AJ, Fiebach JB, Wintermark M, Lindsten A, Smyej J, Bharucha DB, Pedraza S, Rowley HA. Refinement of the magnetic resonance diffusion-perfusion mismatch concept for thrombolytic patient selection: insights from the desmoteplase in acute stroke trials. Stroke. 2012 Sep;43(9):2313-8. doi: 10.1161/STROKEAHA.111.642348. Epub 2012 Jun 26. PMID 22738918
- [Derived] Fiebach JB, Al-Rawi Y, Wintermark M, Furlan AJ, Rowley HA, Lindsten A, Smyej J, Eng P, Warach S, Pedraza S. Vascular occlusion enables selecting acute ischemic stroke patients for treatment with desmoteplase. Stroke. 2012 Jun;43(6):1561-6. doi: 10.1161/STROKEAHA.111.642322. Epub 2012 Apr 3. PMID 22474060
- [Derived] Hacke W, Furlan AJ, Al-Rawi Y, Davalos A, Fiebach JB, Gruber F, Kaste M, Lipka LJ, Pedraza S, Ringleb PA, Rowley HA, Schneider D, Schwamm LH, Leal JS, Sohngen M, Teal PA, Wilhelm-Ogunbiyi K, Wintermark M, Warach S. Intravenous desmoteplase in patients with acute ischaemic stroke selected by MRI perfusion-diffusion weighted imaging or perfusion CT (DIAS-2): a prospective, randomised, double-blind, placebo-controlled study. Lancet Neurol. 2009 Feb;8(2):141-50. doi: 10.1016/S1474-4422(08)70267-9. Epub 2008 Dec 25. PMID 19097942